CLINICAL TRIAL: NCT01633788
Title: A Study of AGN-195263 for the Treatment of Meibomian Gland Dysfunction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 195263-006
Record Dates: First submitted 2012-07-02; First posted 2012-07-04 (Estimated); Results first posted 2017-09-08 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-08

CONDITIONS: Meibomian Gland Dysfunction
MeSH Terms: conditions — Meibomian Gland Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- AGN-195263 0.1% (Experimental): 1 drop of AGN-195263 0.1% instilled in each eye twice daily.
  Interventions: Drug: AGN-195263 0.1%
- AGN-195263 0.03% (Experimental): 1 drop of AGN-195263 0.03% instilled in each eye twice daily.
  Interventions: Drug: AGN-195263 0.03%
- AGN-195263 0.01% (Experimental): 1 drop of AGN-195263 0.01% instilled in each eye twice daily.
  Interventions: Drug: AGN-195263 0.01%
- AGN-195263 Vehicle (Placebo Comparator): 1 drop of AGN-195263 vehicle (placebo) instilled in each eye twice daily.
  Interventions: Drug: AGN-195263 Vehicle

INTERVENTIONS:
Drug: AGN-195263 0.1% — 1 drop of AGN-195263 0.1% instilled in each eye twice daily.
  Arms: AGN-195263 0.1%
Drug: AGN-195263 0.03% — 1 drop of AGN-195263 0.03% instilled in each eye twice daily.
  Arms: AGN-195263 0.03%
Drug: AGN-195263 0.01% — 1 drop of AGN-195263 0.01% instilled in each eye twice daily.
  Arms: AGN-195263 0.01%
Drug: AGN-195263 Vehicle — 1 drop of AGN-195263 vehicle (placebo) instilled in each eye twice daily.
  Arms: AGN-195263 Vehicle

SUMMARY:
This study will evaluate the safety and efficacy of AGN-195263 compared to vehicle in patients with meibomian gland dysfunction (MGD) in the eyelids.

ELIGIBILITY:
Inclusion Criteria:

* Meibomian gland dysfunction in both eyes
* Best-corrected visual acuity of 20/40 or better in each eye

Exclusion Criteria:

* Known or suspected prostate cancer
* History of breast cancer
* Using LATISSE® or any other eye lash growth-stimulating product at least 30 days prior to the screening visit, or anticipated use during the study
* Contact lens wear in either eye during any portion of the study
* Unable to instill eye drops correctly
* History of corneal refractive surgery in either eye within 1 year

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2012-08-22 (Actual); Primary Completion 2015-02-05 (Actual); Study Completion 2015-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (33):
- United States (33):
  - Cornea Consultants of Arizona, Phoenix, Arizona
  - University of Arkansas for Medical, Little Rock, Arkansas
  - Sall Research Medical Center, Artesia, California
  - Orange County Ophthalmology Medical Group, Inc., Garden Grove, California
  - Lugene Eye Institute, Glendale, California
  - Lakeside Vision Center, Irvine, California
  - Scripps Clinic, La Jolla, California
  - North Valley Eye Medical Group, Inc., Mission Hills, California
  - Eye Research Foundation, Newport Beach, California
  - North Bay Eye Associates, Inc., Petaluma, California
  - Centennial Eye Associates, Centennial, Colorado
  - Colorado Eye Associates, PC, Colorado Springs, Colorado
  - Danbury Eye Physicians & Surgeons, PC, Danbury, Connecticut
  - The Eye Associates of Manatee, LLP, Bradenton, Florida
  - Wohl Eye Center, Bloomingdale, Illinois
  - John-Kenyon American Eye Institute, New Albany, Indiana
  - Durrie Vision, Overland Park, Kansas
  - Taustine Eye Center, Louisville, Kentucky
  - Lifelong Vision Foundation, Chesterfield, Missouri
  - Tauber Eye Center, Kansas City, Missouri
  - Ophthalmology Associates, St Louis, Missouri
  - Comprehensive Eye Care, Ltd., Washington, Missouri
  - Northern New Jersey Eye Institute, PA, South Orange, New Jersey
  - Rochester Ophthalmological Group, PC, Rochester, New York
  - Ophthalmic Consultants Long Island, Rockville Centre, New York
  - South Shore Eye Care, LLP, Wantagh, New York
  - Cornerstone Eye Care, High Point, North Carolina
  - Drs. Fine, Hoffman, and Packer, LLC, Eugene, Oregon
  - Vision Center of Texas, PA, Cedar Park, Texas
  - University of Houston, College of Optometry, Houston, Texas
  - Focus Clinical Research, Salt Lake City, Utah
  - Stacy Smith, MD, PC, Salt Lake City, Utah
  - Virginia Eye Consultants, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients from one site were excluded from the modified intent-to-treat analysis population due to compliance issues. Patients from this site who received study treatment were included in the safety population and are reflected in the participant flow.
Period: Overall Study
Arm/Group | AGN-195263 0.1% | AGN-195263 0.03% | AGN-195263 0.01% | AGN-195263 Vehicle
Started | 57 | 58 | 59 | 58
Completed | 50 | 50 | 49 | 45
Not Completed | 7 | 8 | 10 | 13
Not completed — Adverse Event | 1 | 3 | 3 | 3
Not completed — Lost to Follow-up | 2 | 2 | 2 | 0
Not completed — Personal Reasons | 3 | 1 | 1 | 3
Not completed — Protocol Violation | 1 | 0 | 1 | 0
Not completed — Other Reasons | 0 | 2 | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AGN-195263 0.1% | AGN-195263 0.03% | AGN-195263 0.01% | AGN-195263 Vehicle | Total
Number analyzed (Participants) | 57 | 58 | 59 | 58 | 232
Age, Customized [Number; unit: participants]
  40 year to less than 55 years | 17 | 17 | 20 | 19 | 73
  55 years to 65 years | 26 | 24 | 19 | 18 | 87
  over 65 years | 14 | 17 | 20 | 21 | 72
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 39 | 39 | 39 | 156
  Male | 18 | 19 | 20 | 19 | 76

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Meibum Quality Responders in the Study Eye
Description: Meibum quality response is defined as a patient who experiences a reduction ≥ 50% in the number of meibomian glands with a Meibum Quality Score (MQS) of 2 or 3 in the study eye. The MQS is based on Mathers' meibum quality secretion grading 4-point scale where: 0 = Clear excreta or clear with small particles (normal viscosity), 1 = Opaque excreta with normal viscosity, 2 = Opaque excreta with increased viscosity (gel-like), and 3 = Secretions retain shape (or secretions do not express but a toothpaste-like substance can be seen at the opening of the orifice).
Time Frame: Month 6
Population: Modified intent-to-treat: all randomized and treated patients who have values for meibum quality score at randomization, at least one postrandomization visit, and data at the noted time point
Measure: Number; unit: Percentage of Patients
Arm/Group | AGN-195263 0.1% | AGN-195263 0.03% | AGN-195263 0.01% | AGN-195263 Vehicle
Number analyzed (Participants) | 54 | 56 | 53 | 49
Percentage of Patients | 46.3 | 33.9 | 32.1 | 42.9

2. Secondary Outcome: Percentage of Maximum Meibum Quality Score (MMQS) Responders in the Study Eye
Description: The MQS is assessed based on Mathers' meibum quality secretion grading 4-point scale where: 0 = Clear excreta or clear with small particles (normal viscosity), 1 = Opaque excreta with normal viscosity, 2 = Opaque excreta with increased viscosity (gel-like), and 3 = Secretions retain shape (or secretions do not express but a toothpaste-like substance can be seen at the opening of the orifice). MMQS is calculated for each eye as the maximum of the meibum quality scores of the expressible glands within the 6 central glands of the lower eyelids. A patient is considered to be an MMQS responder at a postrandomization visit if the MMQS in the study eye is 0 or 1 (indicating normal viscosity) at that visit.
Time Frame: Month 6
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | AGN-195263 0.1% | AGN-195263 0.03% | AGN-195263 0.01% | AGN-195263 Vehicle
Number analyzed (Participants) | 54 | 56 | 53 | 49
Percentage of Patients | 20.4 | 23.2 | 15.1 | 22.4

3. Secondary Outcome: Percentage of Complete Overall Ocular Discomfort Responders
Description: Ocular symptoms of blurred vision, burning, dryness, eye pain, light sensitivity, itching, and foreign body sensation are assessed by the patient on a 5-point scale ranging from 0 = none to 4 = very severe. A patient is considered a complete overall ocular discomfort responder if the overall ocular discomfort score is 0 (indicating no overall ocular discomfort) at that visit.
Time Frame: Month 6
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | AGN-195263 0.1% | AGN-195263 0.03% | AGN-195263 0.01% | AGN-195263 Vehicle
Number analyzed (Participants) | 55 | 56 | 54 | 51
Percentage of Patients | 20.0 | 19.6 | 14.8 | 9.8

ADVERSE EVENTS:
Description: The Safety Population is used to assess adverse events and serious adverse events and consists of all patients who received at least one dose of study treatment.
Arm/Group | AGN-195263 0.1% | AGN-195263 0.03% | AGN-195263 0.01% | AGN-195263 Vehicle
Serious Adverse Events (participants affected / at risk) | 1/57 | 4/58 | 3/59 | 0/58
Other Adverse Events (participants affected / at risk) | 7/57 | 6/58 | 3/59 | 7/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AGN-195263 0.1% (N=57) | AGN-195263 0.03% (N=58) | AGN-195263 0.01% (N=59) | AGN-195263 Vehicle (N=58)
Gait disturbance (General disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | AGN-195263 0.1% (N=57) | AGN-195263 0.03% (N=58) | AGN-195263 0.01% (N=59) | AGN-195263 Vehicle (N=58)
Eye pruritus (Eye disorders) | 3 | 2 | 2 | 0
Foreign body sensation in eyes (Eye disorders) | 3 | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 3 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 4 | 0 | 1
Prostatic specific antigen increased (Investigations) | 1/18 | 0/19 | 0/20 | 2/19 — Males Only

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.